CLINICAL TRIAL: NCT02653339
Title: Effectiveness of Qufeng Shengshi Fang on Treatment of Allergic Rhinitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS-958
Record Dates: First submitted 2015-12-19; First posted 2016-01-12 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-01

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: traditional Chinese medicine; Loratadine; questionnaire survey
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Loratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Qufeng Shengshi Fang and Loratadine (Experimental): Qufeng Shengshi Fang is a traditional Chinese medicine form 8 kinds of herbs. Loratadine is the second generation antihistamines, after converted into its active metabolite Carrie period (carebastine), its antihistamines and allergy effect has been demonstrated in vitro and in vivo tests, also received data from clinical trials.
  Interventions: Drug: Qufeng Shengshi Fang and Loratadine; Drug: Loratadine
- Loratadine (Active Comparator): Loratadine (INN) is a second-generation H1 histamine antagonist drug used to treat allergies. In structure, it is closely related to tricyclic antidepressants, such as imipramine, and is distantly related to the atypical antipsychotic quetiapine.Loratadine is marketed by Schering-Plough[needs update] under several trade names (e.g., Claritin) and also by Shionogi in Japan. It is available as a generic drug and is marketed for its nonsedating properties. In a version named Claritin-D or Clarinase, it is combined with pseudoephedrine, a decongestant; this makes it useful for colds, as well as allergies but adds potential side effects of insomnia, anxiety, and nervousness.
  Interventions: Drug: Qufeng Shengshi Fang and Loratadine; Drug: Loratadine

INTERVENTIONS:
Drug: Qufeng Shengshi Fang and Loratadine — The patients with allergic rhinitis are divided into two groups, one is experimental group, and the other is control group.
  The experimental group patients are treated with Qufeng by oral, 200ml two times a day and Loratadine by oral,10mg QD
Drug: Loratadine — The patients with allergic rhinitis are divided into two groups, one is experimental group, and the other is control group.
  The control group patients are treated with Loratadine by oral, 10mg QD
  Other Names: Claritin，WS1-(X-014)-2004Z

SUMMARY:
This is a controlled clinical trials about traditional Chinese medicine named Qufeng Shengshi Fang，which consisted of cicada slough，bombyx batryticatus，radix angelicae，radix sileris，honeysuckle flower，forsythia，lithospermum and radix glycyrrhizae，and Loratadine on treatment of Allergic Rhinitis.There are 180 Patients with allergic rhinitis recruited from Department of Allergy and Traditional Chinese.To carry on statistical analysis of the result of the self and between-group cross-reference by two questionnaires filled before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* meet allergic rhinitis (include allergic rhinitis with asthma) diagnostic criteria at Peking Union Medical College Hospital Department of Allergy;
* have allergic rhinitis in episodes.
* without antihistamine,local anaesthetic or traditional Chinese medicine in last months.
* signed the informed consent form.

Exclusion Criteria:

* have severe deviation of nasal septum and nasal polyps.
* have nasal surgery or a history of cancer(tumor).
* have other serious illness or evidence of mental disorders.
* female in pregnancy and lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-03 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Improvement clinical symptoms of Allergen Rhinitis | 0，4 and 8 weeks
  Clinical symptoms of Allergen Rhinitis including Rhinocnesmus (0: No symptom；1：Intermittent；2：Formication but supportable；3：Formication and insupportable)，Sneeze (0: No symptom；1：3-5 times everyday；2：6-10 times everyday；3：>11 times everyday)，Rhinorrhea (0: No symptom；1：modicum；2：medium；3：mass)，Rhinobyon (0: No symptom；1：Conscious inspiratory；2：Intermittent；3：Mostly breathing through mouth)，Itchy eyes(0: No symptom；1：Pruritus but supportable；2：Need rub eyes occasionally；3：Need rub eyes frequently)，Racryorrhea (0: No symptom；1：With sneezing；2：between 1and 3；3：No sneeze also )，Itchy ears and palate(0: No symptom；1：Intermittent；2：Pruritus but supportable；3：Pruritus and insupportable). Assessing the change by comparing the symptom score before and after treatment.

SECONDARY OUTCOMES:
Liver Function Examination | 0，4 and 8 weeks
  Liver function examination including alanine aminotransferase (ALT) (U/L) , aspartate transaminase (AST) (U/L) and glutamyl transpeptidase （GGT）(U/L).
Renal Function Examination | 0，4 and 8 weeks
  Renal function examination including blood urea nitrogen(BUN)（mmol/L）and urine creatinine(UCr) (mmol/d).
Secretory immunoglobulin E Examination | 0 and 8 weeks
Blood Routine Examination | 0，4 and 8 weeks
  Blood Routine Examination including white blood cell(WBC)(*10^9/L),monocyte number（MONO#）(*10^9/L)，monocyte percentage (MONO%)(%)，lymphocyte number（LY#）(*10^9/L)，lymphocyte percentage (LY%)(%)，neutrophil number（NEUT#）(*10^9/L)，neutrophil percentage (NEUT%)(%)，eosinophil number（NEUT#）(*10^9/L)，eosinophil percentage (NEUT%)(%)，red blood cell(RBC)(*10^12/L),hemoglobin(HGB) (g/L) and platelet count(PLT)(*10^9/L).
Urine Routine Examination | 0，4 and 8 weeks
  Urine Routine Examination including occult blood(BLD)(Cells/μL) and proteinuria(PRO)(g/L).
Fractional Exhaled Nitric Oxide Examination | 0 and 8 weeks
Test of Cytokine | 8 weeks
  Cytokines is a kind of low-molecular-weight soluble protein, which has function of regulating inherent immunity and adaptive immunity, erythropoiesis, cell growth and injured tissue repair and others.In the study FlowCellect™ Mouse Th2 Intracellular Cytokine Kit (FCIM025124) and Th17 Intracellular Cytokine Kit (FCIM025125) will be used to compare the change on cytokine before and after treatment. This FlowCellect Mouse Cytokine Th2 Identification Kit for flow cytometry is designed to enable a researcher a quick & easy way to detect IL-4 expression in mouse Th2 CD4+ T-cells. This FlowCellect Mouse Cytokine Th17 Identification Kit for flow cytometry is designed to enable a researcher a quick & easy way to detect IL-17 expression in mouse Th17 CD4+ T-cells.
Test of Metabonomics | 8 weeks
  Metabolomics is the scientific study of chemical processes involving metabolites. Specifically, metabolomics is the "systematic study of the unique chemical fingerprints that specific cellular processes leave behind", the study of their small-molecule metabolite profiles. The metabolome represents the collection of all metabolites in a biological cell, tissue, organ or organism, which are the end products of cellular processes. Small molecules are the objects in Metabonomics which relative molecular mass is less than 1000.In the study NMR will be used as a way to assess the change on Metabonomics before and after treatment.
Test of Proteomics | 8 weeks
  The proteome is the entire set of proteins expressed by a genome, cell, tissue or organism at a certain time. More specifically, it is the set of expressed proteins in a given type of cell or organism, at a given time, under defined conditions. The term is a portmanteau of proteins and genome. Proteomics is the study of the proteome.In the study Mass Spectrometry will be used to compare the change on proteome before and after treatment.
Change of Exosomes | 8 weeks
  Exosomes as a utricle bubble structure are widely distributed in the peripheral blood, urine, saliva, ascites, amniotic fluid, and other body fluids. Exosomes carry different components, which are secreted by different cells, and these components give exosomes a variety in biological functions, such as potential biomarkers of immune cells, cancer, etc.In the study Ribo™ Exosome Isolation Reagent (for plasma or serum) will be used to compare the change on exosomes before and after treatment.
IncRNA Sequencing | 8 weeks
  Long non-coding RNAs (lnc RNAs) are non-protein coding RNA molecules with the sequence longer than 200 nucleotides. They are four times amount as protein coding transcripts and play important roles in diverse cellular regulations. Function identification of these lncRNAs remains challenging although abundant efforts were put in this field. In the study gene expression profile , named RiboArrayTM lncDETECTTM Human Array, will be used which are provided by RiboBio Co., Ltd.
Pulmonary function Examination | 8 weeks
  Pulmonary function Examination including forced expiratory volume in one second(FEV1)(L), forced vital capacity rate of one second(FEV1.0/FVC)(%), maximal mid-expiratory flow velocity(L/s), maximal expiratory flow in 50% vital capacity(L), maximal expiratory flow in 75% vital capacity(L) and peak expiratory flow rate(PEFR)(L/s).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Liang, Doctor, Study Director — Peking Union Medical College Hospital traditional Chinese medicine department
Locations (1):
- Peking Union Medical College Hospital traditional Chinese medicine department, Beijing, Beijing Municipality, China